CLINICAL TRIAL: NCT01467518
Title: A Phase 1, Open-Label, 2-Period Drug Interaction Study to Assess Steady State Plasma Methadone Enantiomer Pharmacokinetics Following Co-Administration of Methadone QD With Dolutegravir (GSK1349572) 50 mg Twice Daily in Opiate-Dependent, HIV Seronegative Adult Subjects.
Brief Title: Methadone-Dolutegravir (DTG - GSK1349572) Drug Interaction Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 115698
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-03

CONDITIONS: Infections, Human Immunodeficiency Virus and Hepatitis
Keywords: methadone; Opiate-dependent
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; Hepatitis | interventions — dolutegravir; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Other): Subjects will be on individualize stable dose of methdaone for 8 days.
  Interventions: Drug: Methadone
- Period 2 (Other): Subjects will be on individualize stable dose of methadone and open label doses of 50mg Dolutegravir (DTG) every 12 hours for 5 days.
  Interventions: Drug: Dolutegravir; Drug: Methadone

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir is an experimental drug in the integrase inhibitor class for the treatment of HIV. Dose of 50mg every 12 hours for 5 days.
  Arms: Period 2
Drug: Methadone — Methadone is a synthetic opioid used in the treatment of opioid dependence. Subjects will be on individualize stabe dose for 8 days.

SUMMARY:
Dolutegravir (DTG, GSK1349572) is an integrase inhibitor that is currently in Phase 3 clinical development for the treatment of HIV infection. As HIV-infected subjects may also be receiving methadone for opioid dependence, an evaluation of the potential interaction between DTG and methadone is warranted. The primary objective of this study is to determine whether concomitant administration of DTG can affect the pharmacokinetics (PK) of methadone. As a secondary endpoint, the PK of DTG will be compared to historical data. This study will be open-label with subjects receiving DTG and stable doses of methadone. The study will be conducted at one center in Canada in adult male and female subjects.

DETAILED DESCRIPTION:
The study is an open label methadone- doltegravir (DTG, GSK1349572) drug interaction study consist of 2 periods. Subjects must be opiate-dependent and are HIV sero-negative and are on stable dose of methadone 14 days prior to pre-screening. After meeting all eligible criterions, subjects will remain on their individual methadone dose for 3 days in period 1. In period 2, subjects will continue on their individual stable dose of methadone and will receive 50 mg DTG every 12 hours for 5 days. Pharmacokinetics will be collected on Day 3 of period 1 and Day 5 of period 2. Safety measurements will be routine chemistry, haematology and urinalysis. Pharmacodynamic parameters for pupillometry and opioid symptom questionnaire will be collected at the same timepoints as for the pharmacokinetics. Subjects will be discharged after the last PK sample has been collected. A follow-up visit will occur 7-14 days after the last dose of study drug. This study will be conducted at one centre in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator feels that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with positive serology for hepatitis B or C may be entered at the discretion of the investigator, if there is no evidence of active disease or hepatic impairment and it is not a new diagnosis.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Subject is enrolled in a methadone maintenance program for at least 12 weeks prior to Period 1, Day 1, and is expected to continue in the program though the duration of this study.
* Subject is receiving a methadone QD regimen that has remained unchanged for 14 days prior to Pre-Screening Visit and the dose is ≤200mg daily.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented (or self reported history) tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow up visit.
* Body weight >/=50 kg for males and >/=45kg for females and BMI within the range 18.0 - 33.0 kg/m2 (inclusive).
* ALT, alkaline phosphatase and bilirubin </=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug screen. Drugs that will be screened for include amphetamines, barbiturates, cocaine, and PCP.
* The subject has a positive pre-study alcohol screen.
* A positive test for HIV antibody.
* Current use of alcohol, which in the investigator's opinion, would compromise subject's safety and/or compliance with the trial procedures, including subjects who are likely to experience withdrawal symptoms upon abstinence.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Subjects using any concurrent prohibited medication. (see Section 9.2, for details on prohibited medications). Use of common medications which are permitted during the study are listed in Section 9.1 (permitted medications).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pomelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 10 days prior to the first dose of study medication.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, lower or upper GI bleeding, inflammatory bowel disease or pancreatitis should be excluded.
* Subject has inadequate venous access.
* History of Gilbert's disease.
* The subject's systolic blood pressure at screening visit is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG as listed in the protocol.
* Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).
* Any clinically significant arrhythmia, any clinically significant conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses>3 seconds, and non-sustained or sustained ventricular tachycardia.
* Heavy smokers (e.g., >20 cigarettes/day) who are unable to abstain for at least 8 hours as required by the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Composite of Methadone Pharmacokinetics | Day 3 (Period 1) and Day 5 (Period 2) at pre-dose, 1, 2, 3, 4. 6, 8, 12, 16, and 24 hours post-dose.
  Steady state total and R-methadone PK measure: AUC (0-t), Cmax and Ct.

SECONDARY OUTCOMES:
Composite of Methadone and DTG Pharmacokinetics | Day 3 (Period 1) and Day 5 (Period 2) at pre-dose, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hrs post-dose for methadone; pre-dose, 1, 2, 3, 4, 6, 8, and 12 hrs post-dose for DTG. Unbound R-methadone at 3 and 24 hours on Day 3 (Period 1) and Day 5 (Period 2).
  Dolutegravir PK: AUC (0-t), Cmax, C0, Ct, Cmin, and CL/F; Steady state total and R-methadone: C0, Cmin and CL/F; Steady state plasma S-methadone: AUC (0-t), Cmax, C0, Ct, Cmin, CL/F; Ratio of S/R-methadone AUC (0-t); Ratio of S/R-methadone AUC (0-t); Steady state plasma unbound R-methadone plasma concentrations.
Adverse Events -Number of participants with adverse events | Pre-screen visit, Day 1 and Day 5 (Period 2)
  Assessed by change from baseline in vital signs (BP and HR), number of subjects with adverse events and toxicity grading of clinical laboratory tests.
Composite of Methadone and DTG Pharmacodynamics | Day 3 (Period 1) and Day 5 (Period 2) at pre-dose, 1, 3, 6, 12, and 24 post-dose.
  Change from baseline in the subject in the overall opiate agonist score and withdrawal score at post-dose and PK concentrations of methadone alone and in combination; Change in the pupillometry parameters from baseline (minimum pupil diameter [CFBmin], pupillometry area over the effect curve [PAOE] and scores at each time point) and PK concentrations of methadone alone and in combination.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Toronto, Ontario, Canada